CLINICAL TRIAL: NCT06313853
Title: Enhancing Triadic Communication About Cognition for Older Adults With Alzheimer's Disease or Related Dementias Facing a Cancer Management Decision
Acronym: COACH-Cog
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Allison Magnuson, Associate Professor of Medicine, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00007068; R01AG077053 (NIH)
Record Dates: First submitted 2024-02-06; First posted 2024-03-15 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Dementia
MeSH Terms: conditions — Neoplasms; Dementia

STUDY DESIGN:
Intervention Model Description: Cluster-randomized
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COACH-Cog Intervention (Experimental): Oncology clinician intervention components: 1) a brief training video, 2) For each patient/care partner dyad that is subsequently enrolled onto the study that the clinician cares for, the oncology clinician will receive the results of the patient's GA with targeted management recommendations for identified GA domain impairments. Patient/Care partner dyad intervention components: 1) Communication coaching session; 2) Patient GA results with management recommendations to consider discussing with the oncology team will be provided to care partners and patients.
  Interventions: Behavioral: COACH-Cog
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: COACH-Cog — Oncology clinician intervention components: 1) a brief training video (completed once during the duration of the study following enrollment and randomization), 2) For each patient/care partner dyad that is subsequently enrolled onto the study that the clinician cares for, the oncology clinician will receive the results of the patient's GA with targeted management recommendations for identified GA domain impairments Patient/Care partner dyad intervention components: 1) Care partners (and patients if able) will participate in a one-time communication coaching session; 2) Patient GA results with management recommendations to consider discussing with the oncology team will be provided to care partners and patients.
  Arms: COACH-Cog Intervention

SUMMARY:
Building upon prior work, the investigator team developed a communication intervention for older adults with ADRD who are considering a decision about cancer management (adapted intervention: COACH-Cog). The investigators hypothesize that for patients with dual diagnoses of ADRD and cancer, COACH-Cog will increase autonomy support of care partners and patients in the decision-making process, leading to greater acknowledgement and support of cognitive concerns and cognitive-related goals, thereby improving goal concordant care. The investigators are conducting a pilot randomized controlled trial (RCT; cluster randomized by physician) including approximately 45 oncology clinicians and 130 patient/care partner dyads evaluating the effect of COACH-Cog on care partner and patient autonomy support, care partner well-being, goal-concordance, and communication.

ELIGIBILITY:
PATIENTS:

Patient Inclusion Criteria:

1. Be age 65 or older
2. Have a clinical diagnosis of Alzheimer's disease or related dementia (ADRD [Alzheimer's disease, vascular dementia, Lewy body dementia, frontotemporal dementia, or dementia of unknown subtype])
3. Have a clinical diagnosis of cancer (any type or stage)
4. Anticipate a potential decision about cancer-related management, as confirmed by the patient's primary medical oncology clinician.
5. Have a care partner willing and able to participate in the study
6. Are able to read and understand English. The communication coaching session will be delivered in English, thus necessitating this requirement.
7. Be able to provide informed consent (as measured by UBACC) or have a Legally Authorized Representative to provide informed consent

Patient Exclusion Criteria:

Patient exclusion criteria: None

CARE PARTNER:

Care partner inclusion criteria:

1. Age 18 or over
2. Able to read and understand spoken English
3. Able to provide informed consent

Care partner exclusion criteria:

None

ONCOLOGY CLINICIAN:

Oncology clinician inclusion criteria:

1. Oncology clinicians affiliated with the Wilmot Cancer Institute
2. Do not intend to move or retire within the next 2 years.

Oncology clinician exclusion criteria:

None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Care Partner: Health Care Climate Questionnaire (HCCQ) | 4-weeks post oncology clinical encounter
  Care Partner autonomy support; score range: 6-42; higher score is better.

SECONDARY OUTCOMES:
Zarit Caregiver Burden Assessment | 4-weeks post-oncology clinical encounter and 3-months post-oncology clinical encounter
  4-Item Measure Care partner well-being: Caregiver burden; total score range 0-16; Higher score is worse burden.
Horton QOL S-subscale | 4-weeks post-oncology clinical encounter and 3-months post-oncology clinical encounter
  11-Item Measure (Subscale Measure) of Care partner well-being: Quality of Life; Total score range 0-11; higher score is worse quality of life.
Care Partner PROMIS Depression | 4-weeks post-oncology clinical encounter and 3-months post-oncology clinical encounter
  Care partner well-being: Depression; score range 4-20; higher score is worse
Care partner PROMIS Anxiety | 4-weeks post-oncology clinical encounter and 3-months post-oncology clinical encounter
  Care partner well-being: Anxiety; score range 4-20; higher score is worse
Care partner: Patient-Centered Communication in Cancer Care (PCC-Ca) | 4-weeks post-oncology clinical encounter and 3-months post-oncology clinical encounter
  Care partner communication; score range 1-5; higher scores are better
Care partner: Health Care Climate Questionnaire - Age (HCCQ-Age) | 4-weeks post-oncology clinical encounter and 3-months post-oncology clinical encounter
  Care partner Age-related autonomy support; score range 0-28; higher scores are worse
Care partner: Qualitative assessment of goal concordance | 3-months post-oncology clinical encounter
  Care partner: Goal concordance; qualitative analysis if goal concordance occurred (yes/no); range 0-130; higher number better
Care partner: Decision Regret Scale | 3-months post-oncology clinical encounter
  Care partner: Decision regret; score range 5-25; higher score is worse

OTHER OUTCOMES:
Patient: Patient-Centered Communication in Cancer Care (PCC-Ca) | 4-weeks post-oncology clinical encounter and 3-months post-oncology clinical encounter
  Patient communication; score range 1-5; higher scores are better
Patient: Health Care Climate Questionnaire (HCCQ) | 4-weeks post-oncology clinical encounter and 3-months post-oncology clinical encounter
  Patient autonomy support; score range: 6-42; higher score is better.
Patient: Health Care Climate Questionnaire - Age (HCCQ-Age) | 4-weeks post-oncology clinical encounter and 3-months post-oncology clinical encounter
  Patient Age-related autonomy support; score range 0-28; higher scores are worse
Patient Decision Regret Scale | 3-months post-oncology clinical encounter
  Patient: Decision regret; score range 5-25; higher score is worse
Physician Decision Regret Scale | 3-months post-oncology clinical encounter
  Physician: Decision regret; score range 5-25; higher score is worse

CONTACTS AND LOCATIONS:
Overall Officials: Allison Magnuson, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Wilmot Cancer Institute, Rochester, New York, United States